CLINICAL TRIAL: NCT00314041
Title: A Randomized, Double-blind, Controlled, Active Comparator, Phase II Study to Assess the Tolerance and Immunogenicity of Conjugate Meningococcal C (MnCC) Vaccine in Infants When Administered in Conjunction With Primary DTP/Hib Vaccination at 2, 3, and 4 Months of Age.
Brief Title: Study Evaluating the Tolerance of Conjugate Meningococcal C Vaccine in Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 6029A1 D110 P500
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Meningitis, Meningococcal
Keywords: Infant; Conjugate vaccine; Meningococcal; Antibody; Immune memory; Health; Meningococcal Vaccines
MeSH Terms: conditions — Meningitis, Meningococcal | interventions — diphtheria-tetanus-pertussis-haemophilus b conjugate vaccine

INTERVENTIONS:
Biological: Meningococcal C
Biological: DTP/Hib

SUMMARY:
Infant phase: To determine the safety of and production of antibodies by a group C meningococcal conjugate vaccine (MnCC), when given at 2, 3, and 4 months of age with routine vaccines.

Booster phase: To compare the safety of and production of antibodies by MnCC with and without MMR and to compare the antibody response to that produced by a low dose of plain polysaccharide vaccine as a way of investigating immune memory

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants 7-10 weeks of age eligible to receive routine immunization

Ages: 7 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240
Dates: Start 1997-06; Primary Completion 1998-04 (Actual); Study Completion 1998-04 (Actual)

PRIMARY OUTCOMES:
Antibody responses to MnCC and concomitant vaccines

SECONDARY OUTCOMES:
Safety and reactogenicity

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For United Kingdom, ukmedinfo@wyeth.com